CLINICAL TRIAL: NCT03049787
Title: The Effectiveness of Traditional Physical Therapy Versus Home Exercise in Conjunction With Glenohumeral and Subacromial Corticosteroid Injection for the Treatment of Shoulder Adhesive Capsulitis
Brief Title: Formal Physical Therapy (PT) vs. Home PT for Adhesive Capsulitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started as the PI was working on another clinical trial.
Sponsor: Boston Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-32842
Record Dates: First submitted 2017-01-07; First posted 2017-02-10 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Adhesive Capsulitis
Keywords: physical therapy; home exercise; adhesive capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home exercise (Experimental): For the home exercise protocol alone arm, subjects will be given an experimental home exercise program and study team will demonstrate the exercises in the clinic and will direct the subjects to perform the exercises 1-2 times daily until symptom resolution.
  Interventions: Other: Home Exercise Protocol
- physical therapy (Active Comparator): Patients will be prescribed routine physical therapy protocol where they will see a physical therapist twice a week and will be instructed by the physical therapist to perform physical therapy exercises at home daily until symptom resolution, as is the routine practice.
  Interventions: Other: Physical Therapy Protocol

INTERVENTIONS:
Other: Home Exercise Protocol — Home exercise therapy protocol given to patient to be completed at home.
  Arms: home exercise
Other: Physical Therapy Protocol — Formal physical therapy protocol to be given to physical therapist working with patient to direct formal intervention along with a home therapy protocol.
  Arms: physical therapy

SUMMARY:
This study aims to evaluate physical therapy (standard of care) and home exercise vs. home exercise alone for the treatment of adhesive capsulitis.

DETAILED DESCRIPTION:
Patients with adhesive capsulitis receive a glenohumeral and subacromial injection routinely for treatment. In addition, the patients are routinely prescribed physical therapy with a home exercise component. The purpose of this study is to evaluate whether home exercise alone is an alternative option to physical therapy. Patients will be approached about the study after they have agreed to receive a glenohumeral and subacromial injection per standard of care for their clinical treatment. The hypothesis being tested is whether home exercise is alone is as beneficial for pain relief, restoration of range of motion, and improvement in shoulder disability from adhesive capsulitis as physical therapy. Additionally sex differences, diabetes mellitus, endocrine, and mental health histories will be noted.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis of Adhesive Capsulitis (limited range of motion)
2. Given glenohumeral and subacromial injection as part of standard care.
3. Capacity to conduct home exercise program or physical therapy (based upon physician judgment, proximity to physical therapy office and as decided by patient)
4. English speaking
5. 18 years of age or greater

Exclusion Criteria:

1. Prior glenohumeral or subacromial corticosteroid injection within 6 months
2. Prior ipsilateral shoulder surgery
3. Current prescription (narcotic) pain medication use
4. Pain disorder (ex. Fibromyalgia, Reflex Sympathetic Dystrophy)
5. Cervical radiculopathy
6. Full-thickness rotator cuff tear
7. Calcific Tendinopathy (past or present)
8. Advanced Stage osteoarthritis as seen on radiograph
9. Past/present ipsilateral shoulder fracture
10. Women that may be pregnant or nursing (self report)

Past/present physical therapy treatment will be documented, but will not be considered an exclusion factor. The reasoning behind this is that the physical therapy likely was not properly targeting the adhesive capsulitis for the patient to arrive in an orthopaedic clinic and is likely at a similar starting point to most other patients regardless of previous physical therapy. All patients currently enrolled in physical therapy will be assigned to either our physical therapy or home exercise program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index(SPADI) | 6 months compared to baseline score
  shoulder pain and disability index to evaluate shoulder pain and function

SECONDARY OUTCOMES:
Change in Range of Motion (ROM) | 6 months compared to baseline score
  evaluate range of motion
Change in Sane Normal and Pain Visual Analogue Score (SANE) | 6 months compared to baseline score
  Subjective shoulder score to determine shoulder pain/function
Change in Mental Health Index- 5 (MHI-5) | 6 months compared to baseline score
  Mental Health Index- 5 to determine patient mental health status
Change in Short Form- 36 (SF-36) | 6 months compared to baseline score
  Short Form Survey- 36 to determine general overall health for patient
Change in Visual Analog Scale Pain (VAS-Pain) | 6 months compared to baseline score
  Visual analog scale- pain to assess shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: Xinning Li, MD, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No